CLINICAL TRIAL: NCT02690246
Title: A Questionnaire Based Study on Symptoms and Treatment Results in Hereditary Hemorrhagic Telangiectasia (HHT)
Brief Title: Symptoms and Treatment Results in Hereditary Hemorrhagic Telangiectasia
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Urban Geisthoff, Prof. Dr. med., University Hospital, Essen
Other Study IDs: University Clinic Essen
Record Dates: First submitted 2016-02-09; First posted 2016-02-24 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Hereditary Haemorrhagic Telangiectasia (HHT)
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with HHT: patients with Hereditary Haemorrhagic Telangiectasia
  Interventions: Other: questionnaire
- control cohort: indirectly only as a control cohort in questionnaire of affected persons

INTERVENTIONS:
Other: questionnaire — a questionnaire based study
  Groups: patients with HHT

SUMMARY:
Hereditary haemorrhagic telangiectasia (HHT), also known as Rendu-Osler-Weber syndrome, is an inherited multisystemic disorder with recurrent epistaxis, mucocutaneous telangiectasia and visceral arteriovenous malformations. The purpose of this study is to provide data about multiple clinical aspects of HHT and responses to treatment. For comparison of some aspects also data of non-affected relatives is collected (second cohort). the questionnaire has been designed primarily for web based entry, but can also be circulated in paper format on request.

DETAILED DESCRIPTION:
Specific aspects include potential consequences from iron deficiency, efficacy and safety of self-packing, effect of female sex hormones, mortality, effects on the immune system.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of Hereditary Haemorrhagic Telangiectasia

Exclusion Criteria:

* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with HHT; Indirectly we accept healthy volunteers only as control cohort in questionnaires of affected persons.
Sampling Method: Non-Probability Sample
Enrollment: 915 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Effect of nasal self-packing to treat epistaxis on the quality of life in patients with HHT measured mainly by Glasgow Benefit Inventory (GBI) | 34 months
  Hereditary Haemorrhagic Telangiectasia is characterised by recurrent epistaxis which can lead to a feeling to lose control. The investigators examine whether the use of high volume low pressure nasal packing is a secure and practical method to improve patients' quality of life.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 34 months

OTHER OUTCOMES:
Number of patients with restless legs syndrome according to a questionnaire including the criteria by Allen et al., Sleep Medicine 4(2003) 101-119 | 34 months
Number of infectious diseases and complications in comparison to healthy spouses | 34 months
Hormonal changes: Change of number of visible telangiectases during menstrual cycle and pregnancy | 34 months

CONTACTS AND LOCATIONS:
Overall Officials: Urban Geisthoff, Prof. Dr., Study Director — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: Undecided